CLINICAL TRIAL: NCT02326896
Title: The New MACOCHA Score Predicts Intubation Failure of Non-anesthesiologist ICU Trainees
Brief Title: MACOCHA Score Predicts Intubation Failure
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Klinik für Kardiologie, Pneumologie und Angiologie, Heinrich-Heine University, Duesseldorf
Other Study IDs: MACOCHA Score
Record Dates: First submitted 2014-12-23; First posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Intubation; Difficult; Intubation; Complication
Keywords: intubation; intensive care unit; MACOCHA Score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Risk factors for difficult intubation are well described in anesthesiology. But intubation in the intensive care unit (ICU) is a challenging issue, associated with severe life-threatening complications. Non-anesthesiologist trainees performing ICU intubation may not fully appreciate the potential difficulty and complications.

Therefore in this retrospective analysis the MACOCHA score will be used to determine difficult intubation in the ICU and predict intubation failure.

ELIGIBILITY:
Inclusion Criteria:

* patients intubated in the ICU
* >18 years of age

Exclusion Criteria:

* <18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients intubated in the ICU
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Intubation complication | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Tienush Rassaf, MD, Principal Investigator — Division of Cardiology, Pulmonary Disease and Vascular Medicine
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany